CLINICAL TRIAL: NCT00092560
Title: Evaluation of the Efficacy and Safety of Fenofibrate and Ezetimibe Coadministration in Patients With Mixed Hyperlipidemia
Brief Title: Two Investigational Drugs in Patients With Mixed Hyperlipidemia (0653-036)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0653-036; 2004_035
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia
Keywords: mixed hyperlipidemia; high cholesterol; high triglycerides
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: fenofibrate monotherapy

SUMMARY:
The purpose of this study is to evaluate the cholesterol lowering effectiveness and safety of two investigational drugs in patients with mixed hyperlipidemia (high cholesterol and high triglycerides).

DETAILED DESCRIPTION:
The duration of treatment is 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol and high triglycerides

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet the additional criteria as required by the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-C vs. fenofibrate for 12 weeks.

SECONDARY OUTCOMES:
All plasma lipid parameters vs. ezetimibe; all non-LDL lipid parameters vs. fenofibrate; safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Farnier M, Freeman MW, Macdonell G, Perevozskaya I, Davies MJ, Mitchel YB, Gumbiner B; Ezetimibe Study Group. Efficacy and safety of the coadministration of ezetimibe with fenofibrate in patients with mixed hyperlipidaemia. Eur Heart J. 2005 May;26(9):897-905. doi: 10.1093/eurheartj/ehi231. Epub 2005 Mar 21. PMID 15781429
- [Derived] Farnier M, Dong Q, Shah A, Johnson-Levonas AO, Brudi P. Low incidence of paradoxical reductions in HDL-C levels in dyslipidemic patients treated with fenofibrate alone or in combination with ezetimibe or ezetimibe/simvastatin. Lipids Health Dis. 2011 Nov 16;10:212. doi: 10.1186/1476-511X-10-212. PMID 22087637